CLINICAL TRIAL: NCT07377786
Title: Prognostic Values of Platelet Indices and Inflammatory Markers in Patients With HELLP Syndrome( Observational Controlled Study)
Brief Title: Study of Prognostic Values of Platelet Indices and Inflammatory Markers in Patients With HELLP Syndrome.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Jaheen Ali, Resident of Anesthesia,surgical Intensive Care, and Pain Management Faculty of Medicine, Sohag University, Sohag University
Other Study IDs: Soh-Med-25-12-9MS
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: HELLP Syndrome
MeSH Terms: conditions — HELLP Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HELLP syndrome group: Pregnant patients diagnosed with HELLP syndrome enrolled prospectively to evaluate platelet indices and inflammatory markers and their prognostic value on maternal and clinical outcomes.
  Interventions: Diagnostic Test: Group I: 30 patients with HELLP syndrome
- Healthy pregnant controlled group: Healthy pregnant women without hypertensive disorders of pregnancy recruited as a control group for comparison.
  Interventions: Diagnostic Test: Group I: 30 patients with HELLP syndrome

INTERVENTIONS:
Diagnostic Test: Group I: 30 patients with HELLP syndrome — All patients will be subjected to the following in ICU through 48 hrs
  Detailed medical history taking:
  Demographic data (age, weight, height, body mass index (BMI). Physical examination (conscious level-vital signs) Type of anesthesia (spinal -general anesthesia) Number of pregnancies, parity, history of previous pregnancies, smoking status, and history of assisted reproductive treatments.
  Laboratory investigations, indices and inflammatory markers:
  will be obtained after delivery, once the patient is admitted to the intensive care unit. Complete blood counts (CBC). Biochemical analyses [such as aspartate aminotransferase (AST), alanine aminotransferase (ALT), lactate dehydrogenase (LDH), albumin ,bilirubin and creatinine]. The indices include platelet count (PC), MPV, PDW, and plateletcrit (PCT), among these, PDW, an indicator of platelet size heterogeneity, is a marker of platelet function. It is being evaluated as a potential indicator for the risk prediction of

SUMMARY:
This study aims to evaluate the prognostic values of platelet indices and inflammatory markers in patients with HELLP syndrome as:- :-Primary outcome To investigate prognostic values of platelet indices and. . inflammatory markers in HELLP syndrome patients as main indices including (NLR-PLR-MPV-PDW and RDW). .

-Secondary outcome. Evaluation complications of HELLP syndrome including. .

* Maternal complication:- eclampsia, disseminated intravascular coagulation (DIC), liver rupture, placental abruption, stroke, and pulmonary or kidney failure. .
* Fetal complication:-intra uterine fetal death(iufd) ,neonate need for admission to NICU , congintal anomalies .assess APGAR score (which assess appearance(skin color)-pulse(heart rate)-Grimace(reflex irritability)- Activity(muscle tone)-Respiratory(breathing efforts) or umblical cord PH<7. .

DETAILED DESCRIPTION:
Hemolysis, elevated liver enzymes, and low platelet count (HELLP) syndrome is a severe complication in the third trimester of pregnancy. First described by Weinstein in 1982(1)

* HELLP syndrome occurs in up to 0.9% of all pregnancies in the third trimester or in the immediate postpartum period (2)

Associated with adverse pregnancy outcomes, the maternal and perinatal mortality rates of HELLP syndrome may reach up to 23.1% and 56.9% respectively, which is life threatening to both the gravida and the fetus(3)

* Usually, patients develop HELLP syndrome before 36 weeks of gestation with vague symptoms such as malaise (90%), right-upper-quadrant pain (90%), nausea, or vomiting(4)

Preeclampsia (PE) constitutes one of the principal reasons for maternal and perinatal morbidity and mortality worldwide. The circumstance typically implicates formerly healthful normotensive women, after 20 weeks of gestation, typically withinside the third trimester, without regarded threat elements or past deliveries. PE can be further complicated with hemolysis and thrombocytopenia, leading to the emergence of HELLP syndrome. Both conditions are classified as hypertensive diseases of pregnancy (HDP), and their pathogenesis has been linked to an excessive maternal inflammatory response, accompanied by enhanced endothelial activation(5)

. The pathogenesis of HELLP is not fully understood. The findings of this multisystem disease are attributed to abnormal vascular tone, vasospasm and coagulation defects. So far, no common precipitating factor has been found. The syndrome seems to be the final manifestation of some insult that leads to microvascular endothelial damage and intravascular platelet activation (6)

* With platelet activation, thromboxane A and serotonin are released, causing vasospasm, platelet agglutination and aggregations, and further endothelial damage. Thus begins a cascade that is only terminated with delivery(7)

Early detection and accurate diagnosis are essential for correct management. The maternal symptoms may be vague and easily mistaken for a variety of medical or obstetric complications which should be excluded. There are two main diagnostic definitions of the HELLP syndrome. The widely used Tennessee classification requires the presence of (1) microangiopathic hemolytic anemia with abnormal blood smear, low serum haptoglobin and elevated LDH levels, (2) elevation of ASAT above 70 IU/L and LD above 600 IU/L (both enzyme levels more than twice the upper limit of normal values) or bilirubin more than 1.2 mg/dL, and (3) a platelet count below 100 109 L1(8) . HELLP syndrome implies impaired placentation during the early stages of pregnancy, associated with hepatic and coagulation cascade involvement. Coagulation system is activated by the contact of platelets with the injured endothelium leading to increase in consumption as well as bone marrow production of platelets. Raised mean platelet volume (MPV) and platelet distribution width (PDW) have been shown to be correlated with severity of the disease, whenever there is decreased PLT count (9)

. The inflammatory reaction in HELLP syndrome is more severe, but studies on the levels of inflammatory indices [e.g., neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), MPV, PDW, monocyte-to-lymphocyte ratio (MLR)] in HELLP patients have rarely been reported. As NLR, calculated by dividing the absolute neutrophil count by the lymphocyte count, reflects the balance between innate (neutrophil-mediated) and adaptive (lymphocyte-mediated) immunity, with elevated values indicating heightened inflammatory activity. PLR, obtained by dividing platelet count by lymphocyte count, integrates the pro-thrombotic and inflammatory roles of platelets with immune regulation. MLR, the ratio of monocytes to lymphocytes, is considered a marker of chronic inflammation and monocyte activation. MPV represents the average size of circulating platelets and serves as an indicator of platelet activation, while PDW measures the variability in platelet size reflecting heterogeneity in platelet production and turnover (10)

. Sisti et al (11, 12)found that the NLR was higher and the PLR was lower in patients with HELLP syndrome in the third trimester, but these indices in the first trimester did not predict the occurrence of HELLP in the third trimester. Only a relatively small number of cases were included in previous studies on this topic and no simultaneous comparison of normal pregnancies and HELLP was found (13, 14)

.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 and 45 years. Gestational age ranged from 28 to 41 weeks. Pregnant women diagnosed with HELLP syndrome. Preeclampsia with Hellp syndrome. Pt with HELLP syndrome was delivered by ceserian section(SC)then admitted to Intensive care unit (ICU) only normal singleton pregnancies without fetal congenital or chromosomal anomalies

Exclusion Criteria:

* Patients with infection and fever. Women with a history of diabetes, hypertension, systemic or endocrine disorder, chronic infection, chronic renal disease Liver diseases. Blood diseases. Drugs affecting platelet counts or functions. Any history of membrane rupture

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — HELlP syndrome in pregnant woman
Study Population: Patients with HELLP syndrome in surgical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
This study aims to evaluate the prognostic values of platelet indices and inflammatory markers in patients with HELLP syndrome | 48Hours
  To investigate prognostic values of platelet indices and. . inflammatory markers in HELLP syndrome patients as main indices including (NLR-PLR-MPV-PDW and RDW)

SECONDARY OUTCOMES:
Evaluation complications of HELLP syndrome | 48 hours
  Maternal complication:- eclampsia, disseminated intravascular coagulation (DIC), liver rupture, placental abruption, stroke, and pulmonary or kidney failure. .
  *Fetal complication:-intra uterine fetal death(iufd) ,neonate need for admission to NICU , congintal anomalies .assess APGAR score (which assess appearance(skin color)-pulse(heart rate)-Grimace(reflex irritability)- Activity(muscle tone)-Respiratory(breathing efforts) or umblical cord PH<7. .

IPD SHARING:
Plan to Share IPD: No